CLINICAL TRIAL: NCT01849510
Title: Efficacy of Dose Intensified Radiotherapy of Spinal Metastases of Solid Tumors by Dose Increased, Homogeneous Radiation of Vertebral Body and Simultaneous Application of Stereotactic Boost.
Brief Title: Efficacy of Dose Intensified Radiotherapy of Spinal Metastases by Hypofractionated Radiation and IGRT hfSRT Mediated Boost
Acronym: SPIN-MET
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPIME2013
Record Dates: First submitted 2013-04-18; First posted 2013-05-08 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Spinal Metastases
Keywords: spinal metastases; vertebral body; stereotaxis; image-guided radiotherapy; hypofractionated; dose intensified; dose elevation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dose intensified (Experimental): hypofractionated 12x3 Gy + integrated boost 12x4 Gy
  Interventions: Radiation: hypofractionated 12x3 Gy + integrated boost 12x4 Gy
- standard (Active Comparator): hypofractionated 10x3 Gy
  Interventions: Radiation: hypofractionated 10x3 Gy

INTERVENTIONS:
Radiation: hypofractionated 12x3 Gy + integrated boost 12x4 Gy — hypofractionated, homogeneous radiation (12x3 Gy) with simultaneously administrated, integrated boost (12x4 Gy) mediated by IGRT & hfSRT
  Arms: dose intensified
Radiation: hypofractionated 10x3 Gy — hypofractionated, homogeneous radiation (10x3 Gy)
  Arms: standard

SUMMARY:
Spinal metastases indicate for an incurable course of disease. Local tumor control after palliative radiotherapy of spinal metastases (10x3 Gy, 1x8Gy) is between 61 to 81%. In 30% of patients, therapy fails locally within two years associated with further symptoms that are difficult to treat, because a further radiation of already radiated vertebra leads to a higher rate of myelitis. This trial aims to improve local tumor control and control of pain by radiotherapy with increase in total and single dose. Dose elevation is realized by simultaneous, integrated boost mediated by image-guided stereotactic radiotherapy (IGRT & hfSRT) and by elevation of elective dose in vertebral body with 12x3 Gy (standard: 10x3 Gy). Primary endpoint is local tumor control (time up to progression). Secondary endpoints are pain control associated with quality of live, severity of acute and chronic adverse effects and overall survival. It is planned to recruit a total number of 155 patients.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18
* expectance of life at least 6 months
* Karnofsky-Score > 50
* 1-3 vertebral body metastases
* Up to 5 other, macroscopic metastases
* effective contraception
* geographic reachability of patients
* Signed study-specific consent form prior to therapy
* no on-treatment participation on other trials

Exclusion Criteria:

* initial required neurosurgical decompression
* rapid, neurological deterioration
* prior radiotherapy of region for planned radiation
* conditions that preclude the application of magnetic resonance tomography
* malignancy: multiple myeloma or lymphoma
* technical conditions preclude stereotactic irradiation (technical limitations of device)
* pregnant or nursing women
* Fertile patients who refuse effective contraception during study treatment
* persistent drug and/or alcohol abuse
* patients that are not able or willing to behave according to study protocol
* absent attendance for personal, disease related data storage and transfer
* on-treatment participation on other trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2013-03; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
tumor control (time up to progression) | up to progression (MR-imaging), max. 5 years after therapy

SECONDARY OUTCOMES:
severity of acute and chronic adverse effects | acute: assessment up to 6 weeks after therapy; chronic: assessment up to 60 months after therapy or up to progression
overall survival | assessment 60 months after therapy or up to death
pain control | assessment 60 months after therapy
  by visual analog scala and questionnaires according pain

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Semrau, MD, Principal Investigator — Strahlenklinik, Universitätsklinikum Erlangen
Locations (3):
- Germany (3):
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Frankfurt; Strahlentherapie, Frankfurt/M.
  - Universitätsklinikum Regensburg, Strahlentherapie, Regensburg